CLINICAL TRIAL: NCT02063347
Title: Innate Human Collateral Supply to Different Vascular Regions
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 185/13; 2451 (Other: University Hospital Berne)
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-07

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: innate collateral supply; collateral; coronary collateral; renal collateral; peripheral collateral; coronary artery disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Coronary artery disease: With coronary artery disease
- No coronary artery disease: Without coronary artery disease

SUMMARY:
Both clinical and experimental studies demonstrate the importance of the pre-existing, ie innate collateral supply in different vascular regions. Furthermore, pathophysiological considerations and experimental data imply an important role for the association of collateral function between different vascular regions.

STUDY HYPOTHESES 1. In the absence of atherosclerotic stenoses, there is a direct association between the collateral function in the coronary, renal and peripheral circulation. 2. The increase in plasma renin in response to a unilateral main renal artery balloon occlusion is inversely related to its functional collateral supply. 3. The decrease in renal vein oxygen saturation in response to a unilateral main renal artery occlusion is inversely related to its functional collateral supply.

DETAILED DESCRIPTION:
Background

PROTECTIVE EFFECT AND INTER-INDIVIDUAL DISTRIBUTION OF THE COLLATERAL CIRCULATION IN DIFFERENT VASCULAR REGIONS

Of all vascular regions, the collateral circulation of the heart is probably the most extensively studied since the initial studies by Fulton.1 The clinical importance of the coronary collateral circulation2 has been established by numerous investigations demonstrating a protective role of well vs. poorly grown coronary collateral arteries.

Whereas involvement of the peripheral arterial network by obstructive arterial disease is frequently asymptomatic, it is, nevertheless, relevant through the association with increased mortality and as a strong predictor of adverse cardiovascular outcomes. The clinical relevance of the collateral circulation in the lower extremities can be epitomized by the discrepancy of frequently encountered long segmental occlusions and the rare occurrence of severe ischemia or amputation. With regard to a systematic evaluation of this apparently well-collateralized region, it was, however, only very recently that assessment using a direct and quantitative method was performed.

Regarding the kidney, the collateral circulation has hitherto been subject to systematic research only in experimental studies,while data in humans are sparse and limited to angiographic assessment. While the hypertensive effect of renal arterial constriction is well-known since the seminal studies of Goldblatt in 1934, the effect of renal collaterals in this context has been neglected despite the readily apparent effects therefrom in the same experiment. The duration of the ensuing hypertension was only short in Goldblatt's experiments with dogs, an observation explained by the abating effect of efficient collaterals on renal artery constriction and consequently developing reduction of the renal ischemia. In humans, only limited and indirect data on the compensatory effect of the renal collateral circulation in the setting of renal arterial constriction exist.The ratio of selective renin concentrations sampled from the renal vein of both kidneys (affected/unaffected) is commonly used to assess the hemodynamic significance of a unilateral renal artery stenosis. Ernst et al., in 37 patients with unilateral renal stenosis, determined the (selective) renal vein renin ratio and additionally performed angiography for presence of renal collaterals( documented in 68%). Renal collaterals tended to normalize renin excretion in a kidney affected by renal artery stenosis. Indeed, 7 patients with a severe stenosis and visible renal collaterals had a normal renin ratio below the cut-off of 1.4. The clinical relevance of renal artery stenosis is underscored by its prevalence in a significant proportion of patients undergoing routine cardiac angiography.22, 23 In the above context, it is noteworthy that hypertension is not present in almost one half of patients with angiographically significant narrowing of a renal artery.

PRE-EXISTING COLLATERAL CIRCULATION AND ITS INTRA-INDIVIDUAL DISTRIBUTION As alluded to before, acute vascular occlusion in arteriosclerosis can ensue in the absence of relevant narrowing. In this situation, solely the native, pre-existing collateral extent can lessen the ischemic tissue injury. On the other hand, the gradual narrowing of a vessel allows development of large arterial anastomoses from pre-existing smaller arterioles in the process known as arteriogenesis. The notion that the pre-existing collateral extent nevertheless remains the basis for the capacity of anastomoses to enlarge is supported by an instructive experimental study by Zbinden et al.: Flow recovery after superficial femoral artery ligation correlated strikingly with the pre-existing collateral extent. Thus, mice with an already high level of pre-existing collaterals had concordantly high flow recovery, while mice with low levels of pre-existing collaterals had low flow recovery.

Given the systemic process of atherosclerosis, the preformed or innate human collateral function in the different vascular regions mentioned before is of interest. On a patient level, this relates to the intra-, as opposed to the inter-individual distribution of the collateral network. While the inter-individual distribution of collateral function in humans has been shown to vary widely also in the absence of vascular narrowings, recent experimental studies in mice have shown that innate collateral extent is shared qualitatively in different tissues. However, in humans, the association between the collateral function in different vascular regions in humans has so far not been investigated.

In conclusion, both clinical and experimental studies demonstrate the importance of the pre-existing, ie innate collateral supply in different vascular regions. Furthermore, pathophysiological considerations and experimental data imply an important role for the association of collateral function between different vascular regions.

Objective

To determine the in vivo prevalence and distribution of functional collateral supply in the coronary, renal and peripheral circulation, and the intra-individual association of collateral function between the different vascular territories. Additionally, the effect of renal collaterals on the response of the kidney to a short bout of ischemia will be investigated.

Methods

DESIGN Prospective, comparative observational study with collateral function measurements in the coronary, renal and superficial femoral artery.

PRIMARY STUDY ENDPOINT Pressure-derived collateral flow index (CFI) SECONDARY STUDY ENDPOINTS Intracoronary ECG ST segment shift during temporary coronary balloon occlusion; plasma renin concentration before, immediately and 10 minutes after main renal artery occlusion, sampled from the suprarenal inferior vena cava ; transcutaneous oxygen tension (tcpO2) as obtained during left superficial femoral artery occlusion from the left anteromedial lower leg.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Referred for elective coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria

* Acute coronary syndrome
* Severe cardiac valve disease
* Congestive heart failure NYHA III-IV
* History of renal disease with normal renal function/ solitary kidney
* Renal (abnormal serum creatinin level) or hepatic failure
* Peripheral artery disease > stage I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients electively referred for coronary angiography in the context of chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Collateral Flow index | At baseline

SECONDARY OUTCOMES:
Intracoronary ST segment elevation | At baseline
Transcutaneous oxygen tension (tcpO2) | At baseline
Plasma renin concentration | Before, immediately after and 10 minutes after main renal artery occlusion
Renal vein oxygen saturation | Before, during and immediately after main renal artery occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD Prof, Principal Investigator — Department of Cardiology, Bern University Hospital, Switzerland
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Stoller M, Seiler C. Intraindividual Variability and Association of Human Collateral Supply to Different Arterial Regions. Am J Cardiol. 2016 Feb 15;117(4):685-690. doi: 10.1016/j.amjcard.2015.11.026. Epub 2015 Dec 2. PMID 26772443